#### STATISTICAL ANALYSIS PLAN

# Intention-to-Treat Analysis for Blood Pressure in Older Adult Women Manuscripts HE-2

Version 1.0 May 25, 2022

# Household air pollution and health: A multi-country LPG stove intervention trial As part of the Household Air Pollution Intervention Network (HAPIN) Trial

Trial Registration: NCT02944682

Protocol Version: HAPIN - Main Study Protocol v14.0 20January2022

Modification History: NA

#### 1. INTRODUCTION

This document contains the intention-to-treat (ITT) statistical analysis plan (SAP) for blood pressure in the older adult women, one of four primary outcomes of the HAPIN trial. This SAP will be posted with the trial registration.

### 1.1. Background and Rationale

Globally, nearly 3 billion people rely on solid fuels for cooking and heating, the vast majority in low- and middle-income countries (LMICs). The resulting household air pollution is the most important environmental risk factor in the 2019 global burden of disease, accounting for an estimated 2.3 million premature deaths annually, largely among women and young children. Previous interventions have provided cleaner biomass-based cookstoves but have failed to reduce exposure to levels that produce meaningful health improvements. There have been no large-scale field trials with liquefied petroleum gas (LPG) cookstoves, likely the cleanest scalable intervention.

This study will provide evidence, including costs and implementation strategies, to inform national and global policies on scaling up LPG stoves among vulnerable populations. Ultimately, this will facilitate deeper policy-level discussions as well as identify requirements for initiating and sustaining household air pollution interventions globally.

## 1.2. HAPIN Study Overview

The aim of the HAPIN study is to conduct a randomized controlled trial of LPG stove and fuel distribution in 3200 households in four LMIC settings (Tamil Nadu, India; Jalapa, Guatemala; Puno, Peru; and Kayonza, Rwanda) to deliver rigorous evidence regarding potential health benefits across the lifespan. Each intervention site will recruit 800 pregnant women (aged 18-<35 years, 9 to <20 weeks gestation), and will randomly assign half their households to receive LPG stoves and an 18-month supply of LPG. Controls will not receive the intervention at the commencement of the trial and are anticipated to continue cooking with solid biomass fuels; they will be compensated for their participation in the study. The mother will be followed along with her child until the child is 1 year old. In households with a second, non-pregnant older adult woman (aged 40 to <80 years) we will also enroll and follow her during the 18-month follow-up period in order to assess cardiopulmonary, metabolic, and cancer outcomes. To optimize intervention use, we will implement behavior change strategies. We will assess cookstove use, conduct repeated personal exposure assessments to HAP (PM<sub>2.5</sub>, black carbon, carbon monoxide), and collect dried blood spots (DBS) and urinary samples for biomarker analysis and biospecimen storage on all participants at multiple time points. The primary outcomes are birth weight, severe pneumonia, and stunting at age 1 year in the child, and blood pressure in the older adult woman.

# 1.3. Study Objectives

The HAPIN study will address the following specific aims: (1) using an intent-to-treat analysis, determine the effect of a randomized LPG stove and fuel intervention on health in four diverse LMIC populations using a common protocol; (2) determine the exposure-response relationships for HAP and health outcomes; and (3) determine relationships between LPG intervention and both targeted and exploratory biomarkers of exposure/health effects.

#### 2. STUDY METHODS

## 2.1. Trial Design

HAPIN is a randomized, 2-arm intervention trial with parallel assignment. Study sites in the four countries (Guatemala, India, Peru, Rwanda) have been selected and evaluated based on activities conducted in the formative research. HAPIN uses a rolling recruitment process whereby each International Research Center (IRC) will enroll 800 pregnant women (one per household) and an additional approximately 120 older adult women (this will vary by IRC) from the same households who meet inclusion/exclusion criteria (Section 4.1). Key characteristics of each study site are given in Table 2 of the HAPIN design publication (Clasen et al. 2020).

Recruitment and enrollment will occur over approximately 15 months at ~53 pregnant women/8 older adult women per month per IRC. All participants will be followed longitudinally for ~18 months (until the child is age 1 year).

#### 2.2. Randomization

To ensure balance between arms, households have been randomly allocated to intervention or control arms as and when they consent to participate. To maintain balance of treatment assignments within each study site at the IRCs, a total of 10 randomization strata are implemented as follows.

- The India IRC randomization list is stratified by the two study sites
- The Peru IRC randomization list is stratified by the six study sites
- Guatemala and Rwanda have one site each.

Separate randomization lists have been generated for each field team conducting randomization at each IRC. Two randomization lists are produced for each of those field teams: one for households that include an older adult woman, and one for households that do not. Additional details on randomization of households can be found in the HAPIN protocol.

## 2.3. Sample Size Considerations

For power calculation for blood pressure, we assume the number of post-randomization to be m=5 and an intraclass correction of p=0.76 for all individuals. The power for detecting a difference in average blood pressure  $(\beta_1)$  in an analysis-of-covariance analysis with baseline blood pressure adjustment for n individuals per arm can be approximated by Frison and Pocock (1992):

$$\Phi\left(-Z_{1-\alpha/2} + \frac{|\beta_1|}{\sqrt{\frac{2\sigma^2}{nm}[1+(m-1)p-mp^2]}}\right).$$

| | Parameter | Sample<br>Size Per<br>Arm | -20% | -10% | Original | +10% | +20% | Previous Studies<br>Estimate (95% CI) |
|---|---|---|---|---|---|---|---|---|
| Change in mean<br>blood pressure<br>(mm Hg) | $\sigma^2$ | 200 | 2.30 | 2.44 | 2.58 | 2.70 | 2.82 | 3.7 (-0.6, 8.1) <sup>a</sup> |

<sup>\*</sup>We examined the impact of power when the key population parameter (residual variance of blood pressure  $\sigma^2 = 12^2$  are set to  $\pm 10\%$  and  $\pm 20\%$  of their values. Calculations assume a 10% attrition during follow-up.

#### 2.4. Trial Framework

HAPIN is a superiority trial. The intention-to-treat analysis is a test to evaluate whether the outcome data are consistent with the assumption of there being no difference between the intervention and control arms.

## 2.5. Statistical Interim Analyses and Stopping Guidance

No interim analysis will be conducted.

## 2.6. Timing of Analysis

All analysis will be conducted once data collection are complete and the SAP has been approved and registered.

## 2.7. Timing of Outcome and Covariate Assessments

Each participating household is to be followed from enrollment until the index child reaches (or would have reached, assuming a live birth and continued vitality) his/her first birthday. For the participating older adult woman in a household the follow up time is approximately 18 months, including baseline measurements (prior to randomization and intervention), when the pregnant woman is at 24-28 and 32-36 weeks of gestation, and when the child is 3 months, 6 months, and 12 months of age (up to 6 total visits).

#### 3. STATISTICAL PRINCIPLES

#### 3.1. Confidence Intervals and P-Values

All confidence intervals will be presented at 95% confidence.

Intention-to-treat analysis of the primary blood pressure outcome (systolic blood pressure) will utilize repeated measures to examine differences in mean blood pressure post-randomization while adjusting for baseline systolic blood pressure; the statistical inference test will be a Wald test at an  $\alpha$ -level of 0.0125. The Bonferroni correction for multiple testing, while conservative, is used to control for family-wise type I error rate to be 0.05 under any dependence structure among the four HAPIN primary outcomes.

Analyses of secondary blood pressure outcomes and subgroup analysis will use an  $\alpha$ -level of 0.05 to identify statistically significance. If the effect modifiers have more than two categories, simultaneous hypothesis tests will be used.

# 3.2. Adherence and Protocol Deviations

All homes in the intervention arm will be equipped with Stove Use Monitoring Systems (SUMS) on their traditional stoves, as well as a subset of approximately 80 homes in the control arm of each IRC. Compliance will be checked every two weeks when SUMS data is downloaded.

Behavioral reinforcements (messages and materials) will be delivered when intervention households show any use of their traditional stoves. We will flag households that are using their traditional stove one or more times over the previous two-week monitoring period. After flagging these households, we will probe members of the

<sup>&</sup>lt;sup>a</sup>McCracken et al. (2007) is a study of 120 older women (>38) from the same randomized trial (RESPIRE), which adjusted for confounders.

participating household to ascertain reasons for non-compliance and intervene as necessary. At all behavioral reinforcement visits, a brief questionnaire will be conducted to identify the barriers to LPG stove use in the household and document the messages and materials used to address those barriers. Once specific reasons/factors are determined, personalized behavior change reinforcements will be delivered.

The intention-to-treat analysis will not consider adherence.

## 3.3. Analysis Populations

For each outcome, the analysis will include all valid outcome measurement (*complete-case*). We define loss to follow-up as any reason that contributes to a missing outcome value, including death of the study participant and withdrawal from study prior to measurement. The same population will be used for exposure-response analyses.

<u>Secondary analysis</u> may use various subsets of the study to examine effect modification.

#### 4. TRIAL POPULATION

## 4.1. Eligibility

Pregnant women will be eligible to participate in the study if they fulfill the following inclusion and exclusion criteria at screening:

#### Inclusion criteria:

- Confirmed pregnancy (hCG positive blood or urine test)
- Aged 18 to <35 years (via self-report)</li>
- Uses biomass stove predominantly
- Lives in study area
- 9 <20 weeks gestation confirmed by ultrasound
- Singleton pregnancy (one fetus)
- Viable fetus with normal fetal heart rate (120-180 beats per minute) at time of ultrasound
- Continued pregnancy at the time of randomization confirmed by self-report
- Agrees to participate with informed consent

#### Exclusion criteria:

- Currently smokes cigarettes or other tobacco products
- Plans to move permanently outside study area in the next 12 months
- Uses LPG stove predominantly, or is likely to use LPG predominantly, in the near future

If two pregnant women live in the same household and are interested in participating, the one with the earliest gestational age will be chosen to participate.

An <u>older adult woman</u> in the same household will be eligible to participate in the study if they fulfill the following inclusion and exclusion criteria at screening:

#### Inclusion criteria:

Aged 40 to <80 years (via self-report)</li>

#### Exclusion criteria:

- Currently smokes cigarettes or other tobacco products
- Pregnant (via self-report)
- Plans to move out of her current household in the next 12 months

 Takes blood pressure medication at enrollment and/or point during follow-up (will be included in sensitivity analysis, below)

If two or more older adult women live in the same household and are interested in participating, one woman will be randomly selected to participate (the one with the next birthday[month and day]).

#### 4.2. Recruitment

The following information will be included in the CONSORT flow diagram. All counts will be reported as total and by IRC.

- Reasons for exclusion when assessed for eligibility
- Participants determined to be ineligible after randomization
- Reasons for exits after randomization
  - Voluntary withdrawal
  - Withdrawn by study team
  - Moved away
- Reasons for exclusion due to missing data

## 4.3. Withdrawal/follow-up

The study will record reasons for exit classified into several categories:

- Not eligible
- Participant voluntary withdrawal
- Withdrawn by study team
- Moved away from study area
- Deceased
- Lost to follow up
- Other

For exits due to eligibility, voluntary withdrawal and withdrawal by study team, several pre-specified reasons will be used, as well as the option to fill in other reasons. The last completed visit will also be recorded. Reasons for withdrawal and loss to follow-up will be ascertained as soon as possible.

## 4.4. Baseline Participant Characteristics

For the ITT analysis, baseline characteristics will be summarized by intervention versus control arms, separately by each IRC as defined by Table 2. Means and standard deviations will be calculated for continuous variables and percentages will be calculated for categorical variables. Missing data will be reported as a separate category.

| Table 2. Baseline characteristics of the older adult women and the household to be reported (including participants randomized and not taking blood pressure medication at any time during follow-up) | | |
|---|---|---|
| Variables | Туре | Definition/Assessment Methods |
| Age (years) | Continuous | Calculated as the date at baseline minus the date of birth. Date at baseline is assigned by the date of visit if not missing. |
| Highest level of education completed | Categorical | <ul> <li>No formal education or some primary school</li> <li>Primary school or some secondary school incomplete</li> <li>Secondary school or vocational or university/college</li> <li>Missing</li> </ul> |
| Body mass index (BMI) | Continuous | BMI calculated as the average weight (kg) divided by the average height squared (m <sup>2</sup> ) |

| Household food insecurity score | Categorical | Categories (corresponding score): • Food secure (0) • Mild (1,2,3) • Moderate (4,5,6) / Severe (7,8) • Missing See <a href="http://www.fao.org/3/as583e/as583e.pdf">http://www.fao.org/3/as583e/as583e.pdf</a> |
|---|---|---|
| Minimum diet diversity | Categorical | Categories (corresponding diet diversity score): Low (< 4) Medium (4-5) High (>5) Missing |
| Number of people who sleep in this house | Continuous | Number of people reported to sleep in the house |
| Second-hand smoking | Categorical | Whether someone in the household other than the older adult woman smokes (smoking of the older adult woman was an exclusion criteria) (yes/no/missing) |
| Assets | Categorical | Responses for each of the following 5 items: TV, radio, mobile phone, bicycle, and bank account. (Yes / No / Missing) |

#### 5. DATA ANALYSIS

In this section we provide the analysis approach for the ITT analysis. The primary outcome is systolic blood pressure. We present the primary analysis along with secondary outcomes, subgroup (effect modification), sensitivity, and additional analyses.

### 5.2. Outcome Definitions

This section describes the outcomes, including data collection approaches and calculations for derived outcomes.

Following the 24-hour exposure assessment period, a nurse or trained field worker measured resting blood pressure in the right arm in triplicate (with at least 2 minutes between measurements) using an automatic monitor (model HEM-907XL; Omron®) at the participant's home. Before starting the measurement, the participant was instructed to sit on a chair in a quiet room for 5 min with legs uncrossed, their back supported by the chair, and their arm supported on a table. The participant also confirmed that she had not smoked, consumed alcohol, or caffeinated beverages (coffee, tea, or Coca-Cola), or cooked using biomass in the past 30 minutes. If she had done any of those activities in the 30 minutes prior to the measurement, she was asked to refrain from doing these activities for 30 minutes before proceeding with the measurements.

A participant with a measured systolic blood pressure  $\geq$  140 mmHg and/or a diastolic blood pressure  $\geq$  90 mmHg was checked again during the same visit. If the same result was observed on two measurements, the participant was referred to the nearest health center or hospital to receive age-appropriate treatment. If a participant had systolic blood pressure < 80 mmHg or diastolic blood pressure < 40 mmHg, she was also referred to the nearest health center or hospital. In analyses, the average of all three blood pressure measurements will be used. Systolic blood pressure values less than 70 mmHg and diastolic blood pressure values less than 35 mmHg will be excluded as implausible.

Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP) and mean arterial pressure is calculated as DBP + (SBP - DBP)/3.

## 5.3. Intention-to-Treat Analysis

The following approach will be used for both primary and secondary blood pressure outcomes. After excluding any women who reported using blood pressure medication at enrollment and/or at any visit, repeated

measurements of blood pressure of the older adult woman will be analyzed using a model to examine differences in mean blood pressure post-randomization, while adjusting for baseline BP. Specifically, let  $y_i$  denote the blood pressure for woman i. The regression model is given by

$$\bar{y}_i^{Post} = \beta_0 + \beta_1 X_i + \beta_2 (y_i^{Base} - \bar{y}^{Base}) + \varepsilon_i$$

where for individual i,  $\bar{y}_i^{Post}$  is the average post-randomization blood pressure measurement,  $X_i$  is an indicator variable (0 for control and 1 for intervention),  $\left(y_i^{Base} - \bar{y}^{Base}\right)$  is the centered baseline measurement of blood pressure, and  $\varepsilon_i \sim N(0, \tau_i^2)$  represents independent Normal error. The parameter of interest  $\beta_1$  captures differences in average blood pressure due to the intervention, accounting for baseline blood pressure A Wald's test will be conducted under the null hypothesis of  $\beta_1 = 0$ .

The variance  $\tau_i^2$  is a function of the number of post-randomization measurements for individual i and the between-measurement correlations. Specifically,  $\tau_i^2$  is given by

$$\tau_i^2 = \frac{\sigma^2}{m_i} \left[ 1 + (m_i - 1)p - m_i p^2 \right]$$

where  $m_i$  is the number of post-randomization measurements,  $\sigma^2$  is the cross-sectional between-individual variance of blood pressure at any time point, p is the intra-class correlation of blood pressure among both baseline and post-randomization measurements. Our primary analysis will assume  $\tau_i^2$  to be constant for all participants. In sensitivity analyses, we will estimate p from a random-intercept model and use weighted least-square to account for heterogenous residual variance  $\tau_i^2$  due to the different number of follow-up measurements across individuals.

Subgroup Analysis. Effect modification analyses will be conducted using interaction terms between the indicator variable for the intervention (study arm, control or intervention) and the effect modifiers. The list of pre-specified subgroup analyses for the ITT analysis is given in Table 3. For each categorized subgroup variable a joint (simultaneous) statistical test (Wald chi-square test for categorical variables; t test for continuous variables) will be conducted to evaluate effect modification.

| Table 3. Definition for variables for subgroup analysis for intention-to-treat analysis | |
|---|---|
| Parameter | Subgroup Definitions |
| Age | Continuous and dichotomous (using median age) |
| International Research Center | Guatemala, India, Peru, Rwanda |
| ВМІ | Continuous and categorical (underweight, less than 18.5 and normal, 18.5-24.9, combined; overweight/obese, 25.0 and above); And also with 3 categories (underweight, normal, overweight/obese). |

Secondary Outcomes: We will evaluate diastolic blood pressure, pulse pressure, mean arterial pressure, and change between baseline and last follow-up measurement (~18 months after baseline, when the child is 1 year old) as secondary outcomes.

Sensitivity Analysis. If imbalance between control and intervention groups for a baseline covariate (Table 2) suggests problems with randomization, and the covariate is a potential confounder, covariate-adjusted effects will be evaluated as a sensitivity analysis. We will also conduct an analysis including women taking blood pressure medication.

Additional Analysis: We will also consider mixed effect models to evaluate changes in blood pressure trajectories with participant-specific random intercepts and random slopes. We will also analyze the difference between baseline and final BP ('change score'). This additional does not include baseline BP as a covariate, and will be of particular importance if there is an imbalance in baseline BP between arms, as in some instances including baseline measurements can introduce bias

Missing Data. Our primary approach to missing outcome data will be a complete-case analysis by excluding participants with a missing baseline blood pressure measurement. All follow-up measurements will be used in the ITT analysis. It is anticipated that missing blood pressure will be balanced between intervention arms.

# 5.4. Analysis Replication Plan

Selected components of the intention-to-treat analysis will be replicated by an independent analyst. Sensitivity analyses will not be replicated.

The replication team will receive the following from the Data Management Core (DMC).

- 1. A cleaned analytic dataset where exclusions have been applied following the CONSORT diagram. The dataset will also include characteristics at baseline and covariates for subgroup analysis.
- 2. A table summarizing characteristics at baseline (overall and by IRC).
- 3. The set of outcomes (primary and secondary) and subgroup analysis to be replicated.

Specific replication tasks include:

- 1. Replicate summary statistics (e.g., mean, standard deviation, percentages, proportion missing) in the baseline characteristic table.
- 2. Replicate intention-to-treat analyses for primary and secondary outcomes according to models specified in Section 5.3.
- 3. Replicate results from subgroup analyses (effect modification) for primary and secondary outcomes